CLINICAL TRIAL: NCT02433782
Title: Physiotherapy Protocol by Myofascial Therapy and Randomized Clinical Study in Patients With Hemophilic Arthropathy
Brief Title: Myofascial Therapy in Patients With Hemophilic Arthropathy
Acronym: He-Fascial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: He-Fascial
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Hemophilia
Keywords: Haemophilia; Arthropathy; Pain; Range of motion; Miofascial techniques
MeSH Terms: conditions — Hemophilia A; Joint Diseases; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Treatment through myofascial therapy for the treatment of pain and restricted mobility in patients with hemophilic arthropathy of the knee and ankle
  Interventions: Other: Myofascial therapy
- Control group (No Intervention): No myofascial intervention. Patients continue their treatment with FVIII or FIX concentrates, normally

INTERVENTIONS:
Other: Myofascial therapy — Maneuver of pressure and sliding over the anterolateral compartment of the leg Maneuver of pressure and sliding on the back of the leg Liberation technique of the popliteal fascia Maneuver of pressure and sliding on the anterior thigh Maneuver of pressure and sliding on the iliotibial tract Maneuver of pressure and sliding on the hamstring muscle region. Induction maneuver of ankle anterior compartment Induction maneuver of knee anterior chamber
  Arms: Experimental group

SUMMARY:
Designing a treatment protocol using myofascial therapy for the treatment of pain and restrictions on mobility in patients with hemophilic arthropathy of the knee and ankle.

Pilot with a small number of patients for assessment the effectiveness and safety of the treatment protocol created.

Randomized clinical trial to assess the effectiveness of treatment with myofascial therapy in patients with hemophilia.

Describe the differences in terms of the dependent variables (range of motion, pain and flexibility) in patients with hemophilia who have carried out the treatment.

Report the relationship between the clinical characteristics of patients and the results obtained after the treatment period.

DETAILED DESCRIPTION:
Phase I pilot study with 5 patients with hemophilia for assessment by myofascial therapy protocol designed for this purpose.

Phase II. Randomized, prospective longitudinal clinical study in patients with hemophilia, to assess the efficacy of an intervention with myofascial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hemophilia A and B.
* Patients older than 18 years.
* Patients with a diagnosis of hemophilic arthropathy of the knee and ankle.
* Patients on prophylactic regimen with FVIII / FIX.

Exclusion Criteria:

* Patients without walking ability.
* Patients with a diagnosis of other congenital coagulopathy (eg von Willebrand disease).
* Patients who have developed antibodies to FVIII / FIX (inhibitors).
* Patients with neurological or cognitive impairments that impede understanding of questionnaires and physical test.
* Patients who have not signed the informed consent document.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding frequency | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Change from number of bleeding during treatment and follow-up period at 1 month

SECONDARY OUTCOMES:
Pain | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Change from joint pain during treatment and follow-up period at 1 month
Joint function | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Change from joint health during treatment and follow-up period at 1 month. Haemophilia Joint Health. Measurement instrument: Score and Gilbert score
Range of motion | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Change from range of movement of ankle and knee during treatment and follow-up period at 1 month. Measurement instrument: universal goniometer with the protocol to measurement for patients with hemophilia

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER MEROÑO-GALLUT, PhD, Study Chair — Universidad Católica San Antonio
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Murcia, Spain